CLINICAL TRIAL: NCT00203762
Title: Effect of the South African Public Sector Antiretroviral Treatment Programme on the Performance of Tuberculosis and Immunization Programmes - A Cluster Controlled (Non-Randomized) Trial
Brief Title: Effect of Public Sector Antiretroviral Treatment Programme on Tuberculosis and Immunization Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Free State Department of Health (Unknown); Medical Research Council, South Africa (Other); Knowledge Translation Programme, University of Toronto (Other); Institute for Clinical Evaluative Sciences (Other); London School of Hygiene and Tropical Medicine (Other); University of the Western Cape (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRC 102770-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2004-03

CONDITIONS: Tuberculosis
Keywords: Pragmatic cluster non-randomized controlled trial; antiretroviral treatment; tuberculosis; childhood immunization; primary care; resource-restricted settings
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Behavioral: Public sector antiretroviral treatment programmes

SUMMARY:
A scale-up of public sector antiretroviral treatment (ART) programmes may divert scarce resources from other priority primary care programmes like tuberculosis and childhood immunization.

The purpose of this study is to compare the performance of tuberculosis (TB) and childhood immunization programmes in primary care facilities participating in the South African national antiretroviral treatment programme with those which have yet to be included in the ART programme.

DETAILED DESCRIPTION:
Large-scale public sector antiretroviral treatment programmes, like those planned for sub-Saharan Africa, will compete for scarce resources, in particular scarce human resources, with other priority primary care programmes like tuberculosis and childhood immunization.

This could lead to impaired performance in other priority programmes like childhood immunization while health workers are distracted by the demands of establishing and maintaining ART programmes. On the other hand, ART provisions may have positive spin-offs for related programmes like improved case detection of tuberculosis among HIV-positive patients seeking ART. The impact of the ART programme on primary healthcare more generally must be weighed against the benefits of providing antiretroviral treatment to those with AIDS.

Comparison: Primary care clinics in the Free State province, South Africa. 15 clinics participating in the first phases of the national ART programme will be compared with 24 clinics which have yet to be included in the national treatment programme. The unit of analysis will be the clinic although the outcome data will be collected from individual patients.

ELIGIBILITY:
Inclusion Criteria:

Clinics:

* Intervention: 15 primary care clinics participating in the first phases of the national antiretroviral treatment programme
* Control: 24 primary care clinics yet to be included in the national antiretroviral treatment programme randomly selected after stratification for health district and ranking of clinic size.

Patients:

* All patients attending tuberculosis and childhood immunization programmes at the above 39 clinics one year before and one year after antiretroviral treatment services commenced in these facilities.

Exclusion Criteria:

Clinics:

* Clinics earmarked for the second year of the rollout of the antiretroviral treatment programme.

Patients:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2003-05; Study Completion 2006-12

PRIMARY OUTCOMES:
TB case detection
TB treatment completion
Measles immunization completed by 18 months

SECONDARY OUTCOMES:
TB cure rate
TB mortality rate
TB treatment failure rate
TB treatment interruption rate
Proportion of TB cases that smear positive

CONTACTS AND LOCATIONS:
Overall Officials: L R Fairall, MBChB, Principal Investigator — University of Cape Town Lung Institute
Locations (1):
- University of Cape Town Lung Institute, Cape Town, Western Cape, South Africa